CLINICAL TRIAL: NCT02464241
Title: Color Vision Tests in Children: Comparison of Standardized and Computer-assisted Examination
Brief Title: Evaluation of Different Color Vision Tests in Children
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2014-0340
Record Dates: First submitted 2015-03-30; First posted 2015-06-08 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Color Perception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- normal control: normal control
  Interventions: Other: only examination
- patients: patients with optic or macular pathology or amblyopia

INTERVENTIONS:
Other: only examination
  Groups: normal control

SUMMARY:
The purpose of this study is to investigate which clinical colour vision assessment fits best for preschool children and school children. The investigators are going to investigate children with a known colour vision affecting ocular disease, as well as healthy children without colour vision deficiency. The goal is to compare the usability and validity of three different clinical tests for colour vision assessment which are already well established in adults but not yet in children.

DETAILED DESCRIPTION:
Colour vision is an important part of the visual perception. There exist hereditary and acquired forms of colour vision deficiency. Hereditary forms affect 8% of males and 0.4% of females. Acquired forms can occur due to diseases which affect the retina, optic nerve or parts of the brain involved in colour vision such as the optic tract or visual cortex. Early diagnosis of colour vision deficiency is especially important in children to provide prompt aid through parents, teachers or other persons taking care. Moreover colour vision deficiency can be an early sign of beginning and progressive ocular diseases.

Colour vision assessment is part of standard clinical testing in ophthalmology. In children, colour vision assessment can be difficult, as most of the tests were developed for adults. The investigators are going to investigate the suitability of some of these tests for children. It is planned to investigate 40 children without colour vision deficiency and 40 children with a known colour vision deficiency. The data collection will take 1 year.

The study involves an ophthalmologic examination and the assessment of 3 different colour vision tests. All examinations are non-invasive, performed once and last in total about 1 to 1.5 hours. The visual acuity will be assessed by eye charts and refraction measurement followed by a slit lamp examination of the front sections of the eye and an optical examination of the eyeground. The three coulour vision tests are part of the standard repertoire of the Institute for ophthalmology of the University hospital of Zürich. Each colour vision test will be performed once as a test run and twice as a study examination. In the first test the child is asked to recognize known geometrical figures and pictures on charts. The second test involves the recognition of colored caps and the third test is a computer-assisted examination where the child should denote the position of a coloured area on the screen.

In the children with a known optical disease there will be performed additionally an optical coherence tomography to quantify the disease based morphological changes of the retinal layers. Therefore the pupils have to be dilated with the application of specific eye drops medication. This can lead to transient decrease of visual acuity for about 2-4 hours. The child should not drive a bicycle during this time interval. The principal of Optical coherence tomography (OCT) is similar to medical ultrasonics. However in OCT, there are used light waves instead of ultrasound waves, which allow an exact examination of the retinal cell layers.

All the examinations performed in this study are standardized procedures at the Institute of Ophthalmology of the University hospital of Zürich. No risks or harms are expected in relation with the planed examinations. No payment will be asked for the study related examinations. Neither for patients nor for their health insurances arise any additional costs related to the participation in this study.

ELIGIBILITY:
Inclusion-Criteria:

* Children at the age of 3-10 years old
* Informed Consent
* Patient group: reduced monocular visual acuity with maculopathy, opticopathy or amblyopia.
* Proband group: no disease with influence on the colour vision, age-related normal visual acuity

Exclusion-Criteria:

* High anomalies of refraction (myopia < -6D, hyperopia > +4D)
* Status post eye surgery
* Medication with suspected influence on the visual perception
* Age below 3 years or beyond 10 years.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 80 children (girls and boys) at the age of 3-10 years without (40 children) or with (40 children) an ocular disease such as maculopathy, opticopathy or amblyopia will be included. Probands and patients are recruited from consultations at the eye clinic of the University hospital of Zürich. The ophthalmologic care is provided independently of the patient's decision whether to participate in the study or not. This decision is the own free will of the patient and his or her parents.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2015-01; Primary Completion 2018-08 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Percentage of correct answers per child per test. | one test performed within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christina Gerth-Kahlert, MD, Principal Investigator — University Hospital Zurich, Division of Ophthalmology
Locations (1):
- University Hospital Zurich, Zurich, Switzerland